CLINICAL TRIAL: NCT04225741
Title: Theory-based Training to Promote Breast Cancer Screening Among Women With Breast Cancer Worries: Randomized Controlled Trial
Brief Title: Theory-based Training to Promote Breast Cancer Screening
Acronym: cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, gnacar, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: gulcin
Record Dates: First submitted 2020-01-09; First posted 2020-01-13 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Breast Cancer; Breast Cancer Female
Keywords: Mammography; Breast self-examination; Early diagnosis
MeSH Terms: conditions — Breast Neoplasms; Breast Self-Examination; Disease | interventions — Sensitivity Training Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- training group (Experimental): The single-session training lasted for approximately 40-45 minutes and was conducted in the training room of Sıtmapınarı family health center, as a suitable environment. The health belief model predicts the determinants of preventive health behaviors and explains inadequate participation in disease prevention and screening programs.22,23 Furthermore, this model not only explains behavior regarding screening, but also evaluates the cognitive factors that facilitate health-promoting behaviors.22-24
  Interventions: Behavioral: Training group
- Control Group (No Intervention): None of the interventions described above were applied to the control group.

INTERVENTIONS:
Behavioral: Training group — The single-session training lasted for approximately 40-45 minutes and was conducted in the training room of Sıtmapınarı family health center, as a suitable environment. The health belief model predicts the determinants of preventive health behaviors and explains inadequate participation in disease prevention and screening programs. Furthermore, this model not only explains behavior regarding screening, but also evaluates the cognitive factors that facilitate health-promoting behaviors.
  Arms: training group

SUMMARY:
BACKGROUND: Breast cancer worries are important determinants in relation to behavior favoring breast cancer screening.

OBJECTIVE: To determine the effect of theory-based training to promote breast cancer screening among women with high and low levels of breast cancer worries.

DESIGN AND SETTING: Randomized controlled trial, conducted in two family health centers.

METHODS: In total, 285 women were recruited. Women with low levels of breast cancer worries were included in the first intervention group (112 women) and the first control group (112 women), while women with high levels of breast cancer worries were included in the second intervention group (37 women) and the second control group (43 women). Theory-based training to promote breast cancer screening was given to intervention groups. The women's willingness to undergo breast cancer screening and breast cancer worry scores were evaluated at 1, 3 and 6 months.

DETAILED DESCRIPTION:
Breast cancer is the most frequent type of cancer and the most common cause of cancer death among gynecological cancers. One in every four women with cancer in the world has breast cancer. The International Cancer Agency reported that there were around 2,088,849 new cases and 626,679 deaths due to breast cancer worldwide in 2018. The incidence of breast cancer is higher in developed countries than in developing countries, but the numbers of deaths due to breast cancer are lower in developed countries than in developing countries.

It is known that breast self-examination, clinical breast examination and mammography play an important role in making an early diagnosis of breast cancer. The uptake rate for mammography performed on a regular basis is low because this is an expensive method, considering that not all individuals have health insurance and public funding is inadequate, especially in developing countries. Hence, breast self-examination (which has no cost) and clinical breast examination (which only has low cost) remain important diagnostic methods. Moreover, during clinical breast examination, healthcare professionals have the opportunity to advise on breast cancer, risk factors, prevention methods and screening methods.

ELIGIBILITY:
Inclusion Criteria:

* The participants included did not have any diagnosis of breast cancer, had not been performing breast self-examination regularly (every month), had not previously had a mammogram, had not previously had a clinical breast examination, were not pregnant or breastfeeding and were literate.

Exclusion Criteria:

* Missing data collection forms.

Ages: 20 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 285 (Actual)
Dates: Start 2015-01-22 (Actual); Primary Completion 2017-08-11 (Actual); Study Completion 2017-08-30 (Actual)

PRIMARY OUTCOMES:
Breast Cancer Worry Scale | 6 months
  Breast Cancer Worry Scale: Lerman et al. developed this three-item scale to measure breast cancer worry levels and their effect on daily activities and mood. Lerman subsequently modified the scale, such that it was extended from breast cancer to general cancer and its number of questions was increased to six. Lerman's six-item cancer worry scale was then modified by Timur Taşhan et al. to measure breast cancer worries alone, and a Turkish validity and reliability study on the BCWS was conducted. Thus, overall, the lowest score that can be obtained is 0, and the highest is 24. A total score of less than 12 denotes a low level of worry regarding cancer, and a total score ≥ 12 indicates a high level of worry.

CONTACTS AND LOCATIONS:
Overall Officials: Gülçin NACAR, Msc, Study Director — Inonu University

REFERENCES:
- [Result] Timur Tashan S, Ucar T, Aksoy Derya Y, Nacar G, Erci B. Validity and Reliability of the Turkish Version of the Modified Breast Cancer Worry Scale. Iran J Public Health. 2018 Nov;47(11):1681-1687. PMID 30581784
- See also: Validity and Reliability of the Turkish Version of the Modified Breast Cancer Worry Scale. — http://www.ncbi.nlm.nih.gov/pubmed/30581784